CLINICAL TRIAL: NCT06430840
Title: Addressing Financial and Social Needs Among Patients With Cancer
Acronym: CAN-ASSIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Chao Family Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Gelareh Sadigh, Associate Professor In Residence, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4937; UCI-24-28 (Other: University of California Irvine IRB)
Record Dates: First submitted 2024-05-19; First posted 2024-05-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Financial Hardship
Keywords: Sleep; Cancer; Financial Hardship; financial education; financial navigation; cost communication
MeSH Terms: conditions — Neoplasms; Financial Stress | interventions — Counseling; Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Enhanced Usual Care (EUC) (Active Comparator): Usual care + pre-screening for financial hardship and social risks
  Interventions: Other: Usual care; Other: Screening for financial and social needs
- Arm B: CostCOM (Experimental): Usual care + two 1-hour phone or video sessions with a remote financial counselor including out-of-pocket cost communication, financial navigation and counseling.
  Interventions: Behavioral: CostCOM (Cost Communication, Financial navigation and counseling); Other: Usual care; Other: Screening for financial and social needs
- Arm C: FinEd (Experimental): Usual care + access to local and national resources including (1) a detailed list of local and national resources for financial navigation, and social needs where patients can self-refer and (2) video and online /printed educational materials to improve financial health literacy
  Interventions: Behavioral: Provision of local and national resources to address financial and social needs; Behavioral: Financial Education; Other: Usual care; Other: Screening for financial and social needs

INTERVENTIONS:
Behavioral: CostCOM (Cost Communication, Financial navigation and counseling) — Patients will receive two 1-hour, phone or video sessions with a remote financial counselor, each session will cover each of these 3 components of CostCOM.
  Out-of-pocket cost communication (OOPC): A review of insurance benefits and education of the patient-specific OOPC for anticipated treatment regimen if any (i.e., medication). The OOPC is provided as a total estimate and will be updated at 3-month session in case of changes in treatment or insurance.
  Financial navigation: Real-time professional guidance to identify financial assistance programs (e.g., co-pay, living expenses) that alleviate costs of care and discuss information to improve insurance coverage.
  Financial counseling: To address the range of patients' financial concerns and enroll patients in financial assistance programs.
  Arms: Arm B: CostCOM
Behavioral: Provision of local and national resources to address financial and social needs — Patients will be provided with a comprehensive list of local resources (in patients' preferred language) in Orange County that can help with food insecurity, ir transportation, as well as contact information for national non-profit organization where patients can self-refer for financial navigation (e.g., Patient Advocate Foundation (PAF)
  Arms: Arm C: FinEd
Behavioral: Financial Education — Patient will receive online and paper educational materials on topics such as health insurance and health insurance literacy, navigating hospitals' price estimator tool.
  Arms: Arm C: FinEd
Other: Usual care — Patients in all arms will receive usual care, which includes routine oncology visits, use of available ancillary staff, and internal or external resources for co-pay assistance or free medication per normal clinic procedures.
Other: Screening for financial and social needs — Patients will be screened for financial hardship and health-related social risks.

SUMMARY:
Financial hardship and health-related social needs (e.g., insecurity about food, housing, transportation, utilities) are common among patients with cancer, resulting in health disparities in cancer outcomes. Our study will test the efficacy of a multicomponent financial navigation and counseling program delivered by a financial navigator (CostCOM), vs. direct patient access to financial education materials and comprehensive list of local resources in the absence of a financial navigator (FinEd) vs. practice usual care among newly diagnosed cancer patients who screen positive for financial hardship and social needs. Investigators anticipate that both CostCOM and FinEd compared to enhanced usual care will improve cost-related cancer care nonadherence, financial worry, health insurance literacy, quality of life and sleep quality and decrease number of missed appointments.

DETAILED DESCRIPTION:
Financial hardship and health-related social needs (HRSNs) (e.g., insecurity about food, housing, transportation, and utilities) are common among patients with cancer, resulting in health disparities in cancer outcomes. Addressing financial hardship and HRSNs can mitigate their damaging health effects, yet screening for them is not the standard clinical practice. There is compelling evidence that out-of-pocket cost (OOPC) communication complemented by financial navigation and counseling delivered by a financial navigator (CostCOM intervention) will decrease financial hardship. However, implementation of this intervention is limited given shortage of financial navigators in many cancer centers. There is also evidence that patients with financial hardship have lower financial health literacy and financial self-efficacy. However, it is not clear whether direct access to local community or national resources and financial education (FinEd intervention) in the absence of financial navigators will meet patient's needs. Investigators propose a 3-arm pilot randomized controlled trial to assess potential efficacy differences in adherence, financial hardship, financial health literacy, quality of life, and sleep between CostCOM vs. FinEd vs. enhanced usual care (EUC) among 90 newly diagnosed cancer patients (1:1 non-metastatic vs. metastatic) who receive systemic or radiation therapy and are screened positive for financial and social needs. Our multidisciplinary team has experience with all facets of the proposed intervention. CostCOM patients will participate in two remote counseling sessions at baseline, and 3 months, and will receive (1) OOPC communication, individualized, patient-specific education of the anticipated medication OOPC; (2) Financial navigation, real-time professional guidance to identify financial assistance programs that will alleviate costs of care and discuss information to improve insurance coverage; and (3) Financial counseling to address the range of patients' financial concerns and enroll patients in financial assistance programs. FinEd patients will receive (1) a comprehensive list of local and national resources where patients can self-refer for financial and social needs; and (2) online and paper financial educational materials on topics such as health insurance and health insurance literacy, and navigating price estimator tools. EUC patients will receive usual care enhanced by screening for financial and social needs. Our goals are to compare the efficacy of CostCOM vs. FinEd vs. EUC at 6 months on (1) patient-reported cost-related cancer care nonadherence (defined as self-reported delay, forgo, stop or change in cancer care due to cost concerns), treatment completion and missed appointments (as obtained via medical record); (2) patient-reported financial worry, material hardship, health insurance literacy, and quality of life; and (3) patient-reported and objectively measured sleep quality using a sleep monitor. The study will support feasibility for a larger trial, and reveal efficacy estimates for potential CostCOM vs. FinEd differences in improving cancer patients' outcomes and approaches for incorporation into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Speak English or Spanish
* 18 years or older
* Were diagnosed with any stage of cancer within the last 120 days
* Getting treatment in University of California Irvine-affiliated oncology clinics
* Have already started treatment like radiation, or cancer medication
* Screen positive for financial hardship or health-related social needs

Exclusion Criteria:

* Patients with indolent cancer undergoing observation alone
* Eastern Cooperative Oncology Group (ECOG) Performance status above 2
* Patients not receiving any cancer-directed therapy
* Patients participating in other therapeutic clinical trials covering the cost of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patients' Cost-Related Cancer Care Non-Adherence | Within 6-months after randomization
  Number of patients who report any incidence during the 6 months (measured at 3, and 6 months) when they self-reports a positive response to any of: (1) delay, (2) forego, (3) stop, or (4) change in cancer prescribed medication due to cost, (5) refuse recommended cancer tests, or (6) skip cancer office visits due to cost.

SECONDARY OUTCOMES:
Patients' Treatment Completion | Within 6-months after randomization
  Number of patients who receive all the prescribed cycle of chemotherapy and/or radiation therapy due within the 6-month study period.
Patients' Missed Appointments | Within 6-months after randomization
  Proportion of treatment appointments or office visits that is marked as cancellation or no show in the absence of chart note advising patient not to show up the appointment.
Patients' Material Financial Hardship | Within 6-months after randomization
  Number of patients who report any incidence during the 6-months (measured 3, and 6 months) with a self-reported positive response to any of the following: (1) home sale, refinance or move to affordable rental, (2) loans, (3) reaching credit limits, and (4) bankruptcy) because of their cancer care, or its treatment
Patients' Financial Worry | Within 6-months after randomization
  Patients level of of financial worry regarding their cancer care will be measured using the Comprehensive Score for Financial Toxicity (COST) 11-item (score 0-44). Higher score= Lower financial worry
Patients' Insurance Literacy | Within 6-months after randomization
  Patients level of health insurance literacy measured by 21 items Health Insurance Literacy Measure (Score range 21-84). Higher score= higher health insurance literacy
Patients' quality of life | Within 6-months after randomization
  Quality of life will be measured using Patient-Reported Outcomes Measurement Information System (PROMIS)-10. T scores will be calculated ranging between 0-100. Higher score= higher quality of life.
Patients' Sleep Quality (Subjective) | Within 6-months after randomization
  Patients quality of sleep will be measured by an Insomnia Severity Index (ISI) that evaluates the severity of patients insomnia symptoms. (score 0-28). The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28).
Patients Sleep Quality (Objective) | Within 6-months after randomization
  Patients total sleep time, sleep efficiency, nighttime awakening, and sleep latency, measured through a sleep ActiGraph

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, Principal Investigator — University of California, Irvine
Locations (6):
- United States (6):
  - UCI Health Cancer Center - Newport, Costa Mesa, California
  - UCI Health Chao Family Comprehensive Cancer Center - Fountain Valley, Fountain Valley, California
  - CHAO Family Comprehensive Cancer Center- Irvine, Irvine, California
  - UCI Health Chao Family Comprehensive Cancer Center - Laguna Hills, Laguna Hills, California
  - UCI Chao Family Comprehensive Cancer Center, Orange, California
  - UCI Health - Yorba Linda, Yorba Linda, California

IPD SHARING:
Plan to Share IPD: No